CLINICAL TRIAL: NCT02432625
Title: Rare Diseases Clinical Research Network Brittle Bone Disease Consortium Longitudinal Study of Osteogenesis Imperfecta
Brief Title: BBD Longitudinal Study of Osteogenesis Imperfecta
Status: Recruiting | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Collaborators: Shriners Hospitals for Children (Other); Hospital for Special Surgery, New York (Other); Children's National Research Institute (Other); Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other); University of California, Los Angeles (Other); Oregon Health and Science University (Other); University of Nebraska (Other); Alfred I. duPont Hospital for Children (Other); University of South Florida (Other); Phoenix Children's Hospital (Other); Marquette University (Other)
Responsible Party: Principal Investigator, Brendan Lee, Professor and Chairman, Baylor College of Medicine
Other Study IDs: H36165
Record Dates: First submitted 2015-04-29; First posted 2015-05-04 (Estimated); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Osteogenesis Imperfecta
Keywords: Osteogenesis Imperfecta; Collagen; Brittle Bone Disorder; Rare Disease Clinical Research Network; COL1A2
MeSH Terms: conditions — Osteogenesis Imperfecta; Brittle Bone Disorder; Osteogenesis Imperfecta, Type V

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Blood
  2. Urine
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Osteogenesis Imperfecta (OI) is a rare disorder of increased bone fragility characterized by fractures with minimal or absent trauma, dentinogenesis imperfecta (DI), and, in adult years, hearing loss. It is seen in both genders and all races. The clinical features of OI represent a continuum varying from perinatal lethality to individuals with severe skeletal deformities, mobility impairments, and very short stature to nearly asymptomatic individuals with a mild predisposition to fractures, normal stature, and normal lifespan. Fractures can occur in any bone, but are most common in the extremities. These disorders can be devastating and progressive and result in deformity, chronic pain, impaired function and loss of quality of life.

The overall goal of this study is to answer specific question about the natural history of brittle bone diseases as defined by molecular etiology and to develop the foundation for prospective clinical studies.

DETAILED DESCRIPTION:
The purpose of this natural history study is to perform a long-term follow-up of a large group of people with osteogenesis imperfecta (OI). The research aims are:

1. To collect natural history data on all individuals enrolled in this longitudinal study. The cause of the brittle bone disease will be compared with things like severity, various features and response to treatments.
2. To determine how often people with type I OI have vertebral compression fractures of the spine.
3. To determine how often people with OI develop scoliosis (curvature of the spine).
4. To determine how often people with OI have problems with teeth alignment and how dental health impacts a person's quality of life.
5. To determine the effect of pregnancy in women with OI.

There will be a total of 1000 people with OI in this study. Participants will be asked to come in every year if 17Y and younger or every other year if 18Y and older for a total of five years.

The following information will be collected at the study visits:

Birth History and past surgical history, Current medical history, Scoliosis evaluation, Walking ability Questionnaire, Dental Quality of Life Questionnaire, Scoliosis and fractures Quality of Life Questionnaires, Physical development evaluation, Medications Use

The following tests will be performed:

Physical exam, dental exam, lung function test, hearing test, mobility test.

The following X-rays will be taken:

DEXA scan, X-ray of the spine, X-ray of the jaw.

Biospecimen (urine and blood) samples will be collected.

ELIGIBILITY:
Natural History Study:

Inclusion Criteria:

* Individuals with OI diagnosed by molecular (DNA) analysis OR
* Individuals whose clinical history and radiographs are highly suggestive of OI, but whose diagnosis has not been verified by biochemical or molecular studies

Exclusion criteria:

* Individuals who are unable to return for their scheduled follow up visits.
* Individuals with skeletal dysplasias other than OI
* Individuals with OI and a second genetic or syndromic diagnosis

Vertebral Compression Fractures component Inclusion criteria

• Patients with nonsense or frameshift mutations in COL1A1 or COL1A2 of any age and clinical features of OI type I.

Exclusion criteria

* Use of a bone-acting treatment agent such as bisphosphonates, calcitonin, calcitriol, fluoride, etc., within one year of enrollment.
* Conditions other than Osteogenesis Imperfecta-HaploInsufficiency (OI-HI) affecting muscle and/or bone development (i.e. cerebral palsy, rickets)
* Nonsense or frame shift mutations in the final coding exons of COL1A1 or COL1A2, as this may not lead to haploinsufficiency.

Scoliosis in OI component:

Inclusion Criteria

* All study participants between the ages of 3 to 17 years OR
* Study participants 18 years and older with scoliosis

Dental and Craniofacial Abnormalities in OI component:

Inclusion Criteria • All subjects aged 3 years and older enrolled in the Longitudinal Study Exclusion Criteria Subjects who refuse the dental examination

Pregnancy in OI component:

Inclusion criteria

• Females of reproductive age with mutations in any known gene causing OI, who are contemplating pregnancy within 5 years of enrollment in the Natural History Study OR Females who are pregnant with available pre-pregnancy BMD (within 5 years prior to the first pregnancy visit).

Exclusion criteria

* Males
* Females who are peri-menopausal or menopausal
* Females who had gestations associated with higher order multiples.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with a diagnosis of Osteogenesis Imperfecta are eligible to enroll in the natural history study.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-06-01 (Actual); Primary Completion 2030-08-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Natural History of OI | 10 years
  The molecular basis of the brittle bone disease will be correlated with phenotype, disease progression and response to current standard of care therapies.

SECONDARY OUTCOMES:
Incidence and progression of scoliosis in OI | 10 years
  Incidence and progression of scoliosis in OI analyzed by subtype and Cobb Angle assessment
Number Vertebral compression fractures in OI HaploInsufficiency | 10 years
  Number and location of Vertebral compression fractures in OI-HI
Incidence of Oral and craniofacial anomalies | 10 years
  Incidence and progression of oral and craniofacial anomalies as captured by panorex and dental exam
Satisfaction of Oral Health 15Y+ | 10 years
  Satisfaction of Oral health as measure by the OHIP 20
Satisfaction of Oral Health 11Y-14Y | 10 years
  Satisfaction of Oral health as measure by the Oral health QOL 11-14Yrs
Effect of pregnancy in women with OI | 10 years
  Change in Spine, Hip, and radius Bone Mineral Density in pregnant women with OI

CONTACTS AND LOCATIONS:
Overall Officials: V. Reid Sutton, M.D., Study Chair — Baylor College of Medicine; Frank Rauch, M.D., Study Chair — McGill University
Locations (12):
- United States (11):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - University of California Los Angeles, Los Angeles, California
  - AI Dupont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of South Florida, Tampa, Florida
  - Kennedy Krieger Institute / Hugo W. Moser Research Institute, Baltimore, Maryland
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hospital for Special Surgery, New York, New York
  - Oregon Health and Science University, Portland, Oregon
  - Baylor College of Medicine, Houston, Texas
  - Shriners Hospital for Children, Chicago / Marquette University, Milwaukee, Wisconsin
- Shriners Hospital for Children, Montreal, Quebec, Canada